CLINICAL TRIAL: NCT02345356
Title: A Randomized, Double-blind Clinical Trial of Anticoagulation Therapy With Warfarin in Caribbean Hispanics: Comparison Between an Admixture-adjusted Pharmacogenetic-driven Warfarin Dose Refinement Algorithm and the Standard of Care
Brief Title: A Genomic Approach to Warfarin Dose Prescription in Admixed Caribbean Hispanics
Status: Completed | Type: Observational
Sponsor: University of Puerto Rico (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Genomas, Inc (Industry)
Responsible Party: Principal Investigator, Jorge Duconge, PhD, MSc, BSc Pharm, Professor, University of Puerto Rico
Other Study IDs: A4070215; 8G12MD007600 (NIH)
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation; Deep Vein Thrombosis; Cardiac Valvular Insufficiency; Coagulopathies; Pulmonary Embolism
Keywords: Pharmacogenomics; Warfarin; Caribbean Hispanics; Polymorphisms; Dosing Algorithm
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Hemostatic Disorders; Pulmonary Embolism | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard-of-Care: the standard clinical approach will be followed
  Interventions: Other: Standard-of-Care
- Genotype-guided: algorithmically guided personalized therapy of warfarin, using a pharmacogenetic model developed in Caribbean Hispanics
  Interventions: Genetic: Genotype-guided

INTERVENTIONS:
Genetic: Genotype-guided — Individual warfarin dose adjustments by using a pharmacogenetically driven algorithm
  Groups: Genotype-guided
Other: Standard-of-Care — Individual warfarin dose adjustments by using a clinically driven algorithm (standard care)
  Groups: Standard-of-Care

SUMMARY:
Caribbean Hispanics are a population with a disproportionately high prevalence of cardio-metabolic disorders but with a limited expectation of benefits from current pharmacogenetic algorithms derived mainly in subjects of relatively pure ancestry. The investigators focus on warfarin responses to develop urgently-needed DNA-driven prescription guidelines for this population, who have arisen from European, West African and Amerindian genomic origins to produce a highly heterogeneous population. Our project combines admixture analysis and DNA-sequencing with development of more accurate rules for better predictability of warfarin dosing to immediately serve this medically underserved population.

DETAILED DESCRIPTION:
Despite the substantial number of work published over the past years in different populations around the world, a fundamental gap remains in understanding whether and how genomic admixture and polymorphisms in warfarin-related pharmacogenes account for the high inter-individual dose variability observed in Caribbean Hispanic patients. In addition to being a medically underserved population, often marginally represented in clinical studies, Caribbean Hispanics are also a genomically heterogeneous population whose high level of admixture has produced a rich repertoire of combinatorial genotypes (e.g., CYP2C9*2/*5 + VKORC1-1639 A/A) that appear to challenge current pharmacogenetic-driven prescribing models. Our project takes a novel approach to definitively assess this admixture component and is also highly practical for its incorporation into a customized pharmacogenetic algorithm that will be implemented in "real-world" clinical settings through a web-based portal. Moreover, the project is also aimed at performing DNA-sequencing to identify those unknown variants on candidate pharmacogenes (i.e., CYP2C9 and VKORC1) that may contribute further to explain dose variability in Caribbean Hispanics. Shaped by strong preliminary data from a SC2 pilot project, the investigators will assess clinical validity and utility of an admixture-adjusted, pharmacogenetic-guided prescribing model for personalized prediction of effective warfarin dosing in Caribbean Hispanics, which also encompasses genetic (common and novel variants) and non-genetic clinical and demographic factors. The study will be conducted over 4 years in 300 patients with thromboembolic disorders receiving warfarin. Four collaborating/recruiting sites will be further connected through precise delivery of genotyping results and prescribing advice to clinicians via a web-based portal. Our novel assessment of genetic admixture will quantify the contribution of European, African and Amerindian ancestry, and the investigators will test whether this admixture component can explain the heritability that is currently missing in the response variability to this drug among Caribbean Hispanics. If successful in our target population, the same approach can ultimately render current pharmacogenomic models for clinical management of related thromboembolic conditions more accurate and predictive for other populations.

The proposed research will advance and expand our understanding of how these clinically relevant variants affect the response to warfarin in an admixed population. Advancing knowledge in the important and under-investigated area of pharmacogenetics in minority populations will generate results that apply to personalize oral anticoagulation therapy in the wider population as it moves, inevitably, toward increasing heterogeneity through admixed genomes.

ELIGIBILITY:
Inclusion Criteria:

* Caribbean Hispanic origin (e.g., Puerto Ricans, Dominicans, Cubans), whose parents are Caribbean Hispanics as well
* Age ≥ 21 years and ≤90 years.
* Willingness and ability to sign informed consent.
* Able to be followed up over 3 months.
* Expected duration of warfarin therapy of at least 3 months.
* Anticoagulation management for the patient will be performed in-hospital and/or as an outpatient by clinicians (i.e., participating Physicians, PharmD) that will adhere to the study dosing algorithms and dose-titration plans.

Exclusion Criteria:

* Non-Hispanic patients (race/ethnicity is self-reported by the patients)
* Age <21 years and >90 years.
* Currently taking warfarin or any other new oral anticoagulant (e.g., Xarelto, Pradaxa, Eliquis, and Savaysa/Lixiana).
* Prior warfarin therapy with known required stable dose.
* Clinician opinion that warfarin dosing needs to be adjusted for reasons not accounted for by dosing algorithm (i.e., other than age, gender, body size, co-meds, comorbidities, diet, genetics, ancestry, INRs and target INR).
* Abnormal baseline INR (off warfarin), e.g., due to liver disease, antiphospholipid antibody
* Contraindication to warfarin treatment for at least 3 months.
* Life expectancy of less than 1 year.
* Pregnant women or childbearing women not using medically approved method of birth control.
* Inability to follow-up on a regular basis with anticoagulation practitioners participating in trial.
* Any factors likely to limit adherence to warfarin, (e.g., dementia, alcohol or substance abuse, plans to move in the next 3 months, history of unreliability in medication taking or appointment keeping, significant concerns about participation in the study from spouse, significant other, or family members, lack of support from primary health care provider).
* Sickle cell, HIV-positive/ AIDS patients
* Cognitive or other causes of inability to provide informed consent or follow study procedures.
* Participating in another trial that prohibits participation in the current trial or planned enrollment in such a trial within the first 3 months of warfarin therapy.
* Anemia: a reduction in Hg ≥2g/dl within 48 hours before randomization and requiring blood transfusions.
* Creatinine Clearance (CrCL) ≤ 15 mL/min.
* Genotype (CYP2C9 or VKORC1) known to participant from prior testing.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caribbean Hispanics (e.g., Puerto Ricans, Dominicans, Cubans), whose parents are Caribbean Hispanics as well.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
time spent within therapeutic range | 6 months
  percentage of time each patient spent within and out of the therapeutic range (TTR) during initiation, using the Rosendaal linear interpolation method.

SECONDARY OUTCOMES:
number of warfarin dose adjustments | 12 weeks
  number of warfarin dose adjustments during the first 12 weeks of therapy
time to stable anticoagulation | 12 weeks
  time to get stabilization of warfarin doses based on achieving at least three consecutive INR measures within the range for the same average dose.
events-free time | 6 months
  the number of days elapsed between warfarin initiation (date of prescription) and the occurrence of the first event of interest. For the purpose of this analysis, we will use a composite of multiple events that includes hospitalization rates (the first hospitalization due to any cause or due to bleeding or thromboembolism), first overanticoagulation (INR> 4) and first major or minor bleeding episode or ischemic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Duconge, PhD, Principal Investigator — University of Puerto Rico Medical Sciences Campus; Graciela M. Vega-Debien, BSc, Study Director — University of Puerto Rico Medical Sciences Campus; Angel Lopez-Candales, MD, Study Director — University of Puerto Rico Medical Sciences Campus; Alga S. Ramos, PharmD, Study Chair — Miami VA Hospital
Locations (3):
- Miami VA Healthcare System, Miami, Florida, United States
- Puerto Rico (2):
  - UPR University Hospital at Carolina, Carolina
  - UDH University Hospital at Centro Medico, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan is fully described in the corresponding section of the protocol. A thorough description of appropriate use of the data to be shared in this study is provided in informed consent documents. Limitations on data use are also described therein and in this Institutional Certification. Safeguards to protect the data according to Federal standards for information protection will be implemented. As stated by guidelines, data will be made available in the database of Genotype and Phenotype (dbGaP) http://www.ncbi.nlm.nih.gov/gap through controlled-access. This research involves individual-level human data. We expect to share both genotypes and phenotype data as well as additional information necessary to interpret such data, and we propose a data sharing plan that complies with NIH guidelines for NIH-funded studies (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-07-088.html) and the new NIH Genomic Data Sharing (GDS) Policy's scope (http://gds.nih.gov/03policy2.html).

REFERENCES:
- [Background] Claudio-Campos K, Duconge J, Cadilla CL, Ruano G. Pharmacogenetics of drug-metabolizing enzymes in US Hispanics. Drug Metab Pers Ther. 2015 Jun;30(2):87-105. doi: 10.1515/dmdi-2014-0023. PMID 25431893
- [Background] Claudio-Campos K, Orengo-Mercado C, Renta JY, Peguero M, Garcia R, Hernandez G, Corey S, Cadilla CL, Duconge J. Pharmacogenetics of healthy volunteers in Puerto Rico. Drug Metab Pers Ther. 2015 Dec;30(4):239-49. doi: 10.1515/dmpt-2015-0021. PMID 26501165
- [Background] Duconge J, Cadilla CL, Seip RL, Ruano G. Why admixture matters in genetically-guided therapy: missed targets in the COAG and EU-PACT trials. P R Health Sci J. 2015 Sep;34(3):175-7. No abstract available. PMID 26454897
- [Background] Duconge J, Ramos AS, Claudio-Campos K, Rivera-Miranda G, Bermudez-Bosch L, Renta JY, Cadilla CL, Cruz I, Feliu JF, Vergara C, Ruano G. A Novel Admixture-Based Pharmacogenetic Approach to Refine Warfarin Dosing in Caribbean Hispanics. PLoS One. 2016 Jan 8;11(1):e0145480. doi: 10.1371/journal.pone.0145480. eCollection 2016. PMID 26745506
- [Result] Claudio-Campos K, Labastida A, Ramos A, Gaedigk A, Renta-Torres J, Padilla D, Rivera-Miranda G, Scott SA, Ruano G, Cadilla CL, Duconge-Soler J. Warfarin Anticoagulation Therapy in Caribbean Hispanics of Puerto Rico: A Candidate Gene Association Study. Front Pharmacol. 2017 Jun 7;8:347. doi: 10.3389/fphar.2017.00347. eCollection 2017. PMID 28638342